CLINICAL TRIAL: NCT00983645
Title: A Prospective, Open-label, Randomized Trial Comparing Prograf and Neoral Use in Kidney Transplant Recipients of Hispanic Ethnicity
Brief Title: A Trial Comparing Prograf and Neoral Use in Kidney Transplant Recipients of Hispanic Ethnicity
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient funding
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 53271
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Results first posted 2015-10-20 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-04

CONDITIONS: Renal Transplant Rejection
Keywords: Kidney Transplantation; Immunosuppression
MeSH Terms: interventions — Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neoral (Active Comparator): Neoral is a pill indicated for the prophylaxis of organ rejection in kidney transplants
  Interventions: Drug: Neoral
- Prograf (Active Comparator): Prograf is a medication used for the prophylaxis of rejection in allogeneic kidney transplants and may be used concomitantly with adrenal corticosteroids.
  Interventions: Drug: Prograf

INTERVENTIONS:
Drug: Prograf — Tacrolimus (Prograf) starting dose 0.05-0.15 mg/kg PO BID
  Other Names: Tacrolimus
  Arms: Prograf
Drug: Neoral — Cyclosporine (Neoral) starting dose 3mg/kg PO BID
  Other Names: Cyclosporine
  Arms: Neoral

SUMMARY:
This study aims to compare outcomes in renal transplant recipients in the hispanic population based on their immunosuppressant regimens.

DETAILED DESCRIPTION:
This study aims to include Hispanics who have undergone a renal transplant to determine the specific outcome after renal transplantation, assuming that ethnic groups require different immunosuppressant regimens. Trough levels in transplant recipients determine the dosing requirements for Tacrolimus and Cyclosproine. It has been recently found, however, that testing cyclosporine levels in the blood 2 hours after taking cyclosporine is more effective in dosing cyclosprine for renal transplant patients than trough levels. The specific study aims include comparing the cyclosporine monitoring in patients with trough and C2 levels, and adjusting immunosuppression based on C2 levels.

ELIGIBILITY:
Inclusion Criteria:

* Cadaveric or Living Donors
* 18 years old or greater
* Primary renal transplants
* Hispanic ethnicity

Exclusion Criteria:

* Prior renal transplant
* Multi-organ transplant
* Recipient with history of Diabetes Mellitus
* PRA > 20%
* Cold Ischemia Time > 24 hours

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-10; Primary Completion 2012-10 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Baron, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Neylan JF. Racial differences in renal transplantation after immunosuppression with tacrolimus versus cyclosporine. FK506 Kidney Transplant Study Group. Transplantation. 1998 Feb 27;65(4):515-23. doi: 10.1097/00007890-199802270-00011. PMID 9500626
- [Background] First MR, Gerber DA, Hariharan S, Kaufman DB, Shapiro R. Posttransplant diabetes mellitus in kidney allograft recipients: incidence, risk factors, and management. Transplantation. 2002 Feb 15;73(3):379-86. doi: 10.1097/00007890-200202150-00011. PMID 11884934
- [Background] Jindal RM, Hjelmesaeth J. Impact and management of posttransplant diabetes mellitus. Transplantation. 2000 Dec 15;70(11 Suppl):SS58-63. No abstract available. PMID 11152233
- [Background] Knoll GA, Bell RC. Tacrolimus versus cyclosporin for immunosuppression in renal transplantation: meta-analysis of randomised trials. BMJ. 1999 Apr 24;318(7191):1104-7. doi: 10.1136/bmj.318.7191.1104. PMID 10213717
- [Background] Pirsch JD, Miller J, Deierhoi MH, Vincenti F, Filo RS. A comparison of tacrolimus (FK506) and cyclosporine for immunosuppression after cadaveric renal transplantation. FK506 Kidney Transplant Study Group. Transplantation. 1997 Apr 15;63(7):977-83. doi: 10.1097/00007890-199704150-00013. PMID 9112351

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neoral | Prograf
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neoral | Prograf | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Full Range); unit: years] | 29.875 [18 to 53] | 42.14 [29 to 56] | 35.6 [18 to 56]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 7 | 15
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 4 | 10
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Rejection
Time Frame: 6 months post-transplant
Population: Data cannot be located for analysis.
Arm/Group | Neoral | Prograf
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Renal Function
Time Frame: 6 months post-transplant
Population: Data cannot be located for analysis.
Arm/Group | Neoral | Prograf
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Post-transplant Diabetes Mellitus
Time Frame: 6 months post-transplant
Population: Data cannot be located for analysis.
Arm/Group | Neoral | Prograf
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Lipid Levels
Time Frame: 6 months post-transplant
Population: Data cannot be located for analysis.
Arm/Group | Neoral | Prograf
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: Standard practice
Arm/Group | Neoral | Prograf
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

LIMITATIONS AND CAVEATS:
A limitation to this study is early termination leading to a small number of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes